CLINICAL TRIAL: NCT06671236
Title: An Open, Single-Arm, Multi-Center Clinical Study to Evaluate the Safety and Tolerability of Regulatory T Cells (Tregs) In the Treatment of Neurodegenerative Diseases
Brief Title: Clinical Study of Regulatory T Cells (Tregs) in the Treatment of Neurodegenerative Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novabio Therapeutics (Industry)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NP001-NDD02
Record Dates: First submitted 2024-10-29; First posted 2024-11-04 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Treg; regulatory T cells; neurodegenerative diseases; Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous Human Polyclonal Regulatory T Cells Injection (NP001 Cell Injection) (Experimental): Regulatory T cell therapy, intrathecal injection
  Interventions: Biological: Autologous Human Polyclonal Regulatory T Cells Injection (NP001 Cell Injection)

INTERVENTIONS:
Biological: Autologous Human Polyclonal Regulatory T Cells Injection (NP001 Cell Injection) — Regulatory T cell therapy, intrathecal injection

SUMMARY:
An open, multi- center phase Ⅰ clinical study evaluating the safety and efficacy of autologous human polyclonal regulatory T cell injection (NP001 cell injection) in patients with Neurodegenerative diseases (ALS).

DETAILED DESCRIPTION:
This is an open-label, non-randomized, multi-center clinical trial of single-agent NP001 cell injection in patients with with Neurodegenerative diseases (ALS).

After subject consents to the study, an apheresis procedure will be performed to collect cells to manufacture the investigational product, NP001 cell injection. NP001 cell injection are manufactured ex vivo to yield enriched Tregs.

This study is evaluating NP001 cell injection at the dose of 1x E6 cells, 1x E7 cells, and 1x E8 cells/times, with up to 3 times separated by 4 weeks among dosing (intrathecally on Days 1, 29, and 57). Study subjects are then followed for several months to capture safety and efficacy parameters. The total duration of NP001 cell injection and follow-up interval on this protocol is approximately 12-months.

ELIGIBILITY:
Inclusion Criteria:

-

Patients must meet all of the following criteria to be eligible for enrollment in this study:

1. Male or female patients aged 18 to 70 years;
2. According to current international diagnostic criteria:

   ALS: defined by the Gold Coast Diagnostic Criteria (Shefner, 2020) as having a diagnosis of sporadic or familial amyotrophic lateral sclerosis (ALS), diagnosed as a probable, probable, or definite patient with laboratory support according to the World Federation of Neurology El Escorial criteria;
3. If there is a stable dose for more than one month prior to study entry. For example, patients with ALS can continue treatment with riluzole (Rilutek®) and/or edaravone (Radicava®);
4. Patients must have > two weeks after the end of major surgery and after the completion of participation in other research trials;
5. Patients must have recovered from clinical toxicity (CTCAE [5th Edition] toxicity values have resolved to < 2);
6. Serum creatinine less than or equal to 2.0 mg/dL;
7. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x upper limit of normal;
8. Bilirubin < 1.5 (except Gilbert's disease);
9. Lung slow vital capacity (SVC) > 70% of predicted normal;
10. No history of abnormal bleeding tendency;
11. Informed consent must be obtained prior to performing any study-related procedures that are not part of standard medical care, with the understanding that the participant may withdraw from the study without influence for the future medical care.

Exclusion Criteria:

-

Subjects with any of the following cannot be enrolled in this study:

1. uncontrolled infection;
2. < 3 drugs do not adequately control hypertension;
3. Documented history of pulmonary embolism within 6 months of enrollment;
4. Clinically significant cardiology, defined as: myocardial infarction, NYHA-graded class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmia, or ECG evidence of acute ischemia or abnormal conduction system within 6 months prior to enrollment;
5. Patients with a history of coronary artery bypass grafting or angioplasty will be evaluated by cardiology and considered on a case-by-case basis;
6. Seropositive for HIV, hepatitis B or hepatitis C;
7. Pregnant or lactating patients;
8. Patients of childbearing potential or males with partners of childbearing potential who are unwilling to use contraception;
9. Participation in any other interventional study;
10. Treatment with another investigational drug, biologic, or device within 30 days or 5 half-lives (whichever is longer) of the screening period. Patient participation in observational/non-interventional clinical studies will be discussed with the Medical Monitor;
11. Prior treatment with ALS gene or cell therapy;
12. History of clinically significant tumor, liver or kidney disease, or other uncontrolled disease;
13. presence of a feeding tube;
14. Current use of antipsychotics, antiepileptic drugs (except benzodiazepines, gabapentin, pre-Bahrain) or class 1 (e.g., flecainide) or class 3 (e.g., amiodarone) antiarrhythmic drugs;
15. Subjects who, in the opinion of the investigator, are at significant risk of suicide;
16. Other conditions that the investigator considers unsuitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Related adverse events (AEs) | 6 months
  Incidence of Treatment Related AEs, AEs of special interest and serious adverse events (SAEs)
Identification of Maximum Tolerated Dose (MTD) | 28 days
  Incidence of dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Amyotrophic lateral sclerosis functional rating scale- revised (ALSFRS-R) | 1 year
  The ALSFRS-R is a simple, validated, and reliable tool for evaluating declines in function. It involves self-rating by patients on their ability and independence across 12 functional activities, with each question scored from 0 to 4 (4 means normal). The total score ranges from 0 (worst) to 48 (best), covering aspects of speech, swallowing, fine motor skills, gross motor skills, and respiratory function.
Rasch Overall ALS Disability Scale (ROADS) | 1 year
  ROADS is a patient-reported outcome measure that assesses overall disability level in patients with ALS. The scale contains 28 items, each scored 0, 1, or 2.
  The scale was constructed and validated using Rasch analyses - a modern test theory technique that produces linearly-weighted scales, meaning that a 1-point change is a quantifiable, consistent measurement of disability across the scale, and a 2-point change reflects twice the amount of disability.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes